CLINICAL TRIAL: NCT06784063
Title: Evaluation of the Impact of Residual Astigmatism on the Visual Performance With Clareon Vivity
Brief Title: Visual Performance With Clareon® Vivity® Intraocular Lenses (IOLs)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILE632-C003
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Astigmatism
Keywords: Cataract; IOL
MeSH Terms: conditions — Astigmatism; Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Clareon Vivity/Vivity Toric (Experimental): Previous implantation in both eyes with Clareon Vivity/Vivity Toric Extended Vision IOLs, with previous implantation defined as at least 4 months prior to study participation.
  Interventions: Device: Clareon Vivity Extended Vision IOL

INTERVENTIONS:
Device: Clareon Vivity Extended Vision IOL — Extended vision intraocular lens implanted in the capsular bag of the eye during cataract surgery. IOLs are intended for long term use over the lifetime of the cataract patient.
  Other Names: Models CNWET0, CNWET3, CNWET4, CNWET5, CNWET6, CNAET0, CNAET3, CNAET4, CNAET5, CNAET6, CCWET0, CCWET3, CCWET4, CCWET5, CCWET6, CCAET0, CCAET3, CCAET4, CCAET5, CCAET6.; Clareon Vivity™ Extended Vision Hydrophobic IOL; Clareon Vivity™ Extended Vision Hydrophobic Toric IOL; Clareon Vivity™ UV Absorbing IOL

SUMMARY:
The purpose of this study is to generate clinical data to quantify the impact of residual astigmatism on the overall visual performance during distance, intermediate, and near viewing in patients implanted with Clareon Vivity IOLs.

DETAILED DESCRIPTION:
This single visit study is designed to help understand how vision is affected if the eye still has astigmatism after cataract surgery. Participants will be individuals who have already undergone cataract surgery and received a Clareon Vivity IOL in both eyes at least 4 months prior to study enrollment. During the study visit, trial lenses (glass lenses that are used during an eye exam) will be used to temporarily create the effect of astigmatism on the eye.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign an Institution Review Board-approved informed consent form;
* Willing and able to attend all scheduled study visits as required by the protocol;
* Implanted with study IOLs in both eyes at least 4 months prior to study participation;
* BCDVA of 0 logMAR or better in each eye.

Exclusion Criteria:

* Residual astigmatism greater than or equal to 1.00 D;
* Clinically significant ocular conditions as specified in the protocol;
* History of ocular surgeries other than limbal relaxing incisions
* Other protocol-specified exclusion criteria may apply.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Mean difference in monocular Best Corrected Distance Visual Acuity (BCDVA) (4 meters) before and after inducing 1.0 diopter (D) astigmatism - WTR | Day 0, coinciding with IOL implantation at least 4 months prior to visit
  BCDVA will be assessed with best refractive correction in place at a distance of 4 meters (m) using Early Treatment Diabetic Retinopathy Study (ETDRS) letter charts. Trial lenses will be used to induce 1.0 diopter (D) of astigmatism with-the-rule (WTR), defined as -0.50/+1.00 D at approximately 180 degrees on the optical axis. VA will be measured in logarithm minimum angle of resolution (logMAR), with a lower logMAR value indicating better visual acuity. The change in VA before and after inducing astigmatism will be reported. One eye (first implanted eye) will be assessed. This is a co-primary endpoint.
Mean difference in monocular Distance Corrected Intermediate Visual Acuity (DCIVA) (66 centimeters) before and after inducing 1.0 D astigmatism - WTR | Day 0, coinciding with IOL implantation at least 4 months prior to visit
  DCIVA will be assessed with distance correction in place (plus or minus power) at a distance of 66 cm from the spectacle plane using ETDRS letter charts. Trial lenses will be used to induce 1.0 D of astigmatism WTR, defined as -0.50/+1.00 D at approximately 180 degrees on the optical axis. VA will be measured in logMAR, with a lower logMAR value indicating better visual acuity. The change in VA before and after inducing astigmatism will be reported. One eye (first implanted eye) will be assessed. This is a co-primary endpoint.
Mean difference in monocular Distance Corrected Near Visual Acuity (DCNVA) (40 cm) before and after inducing 1.0 D astigmatism - WTR | Day 0, coinciding with IOL implantation at least 4 months prior to visit
  DCNVA will be assessed with distance correction in place (plus or minus power) at a distance of 40 cm from the spectacle plane using ETDRS letter charts. Trial lenses will be used to induce 1.0 D of astigmatism WTR, defined as -0.50/+1.00 D at approximately 180 degrees on the optical axis. VA will be measured in logMAR, with a lower logMAR value indicating better visual acuity. The change in VA before and after inducing astigmatism will be reported. One eye (first implanted eye) will be assessed. This is a co-primary endpoint.
Mean difference in monocular Best Corrected Distance Visual Acuity (BCDVA) (4 meters) before and after inducing 1.0 diopter (D) astigmatism - ATR | Day 0, coinciding with IOL implantation at least 4 months prior to visit
  BCDVA will be assessed with best refractive correction in place at a distance of 4 m using ETDRS letter charts. Trial lenses will be used to induce 1.0 D of astigmatism against the rule (ATR), defined as -0.50/+1.00 D at approximately 90 degrees on the optical axis. VA will be measured in logMAR, with a lower logMAR value indicating better visual acuity. The change in VA before and after inducing astigmatism will be reported. One eye (first implanted eye) will be assessed. This is a co-primary endpoint.
Mean difference in monocular Distance Corrected Intermediate Visual Acuity (DCIVA) (66 centimeters) before and after inducing 1.0 D astigmatism.- ATR | Day 0, coinciding with IOL implantation at least 4 months prior to visit
  DCIVA will be assessed with distance correction in place (plus or minus power) at a distance of 66 cm from the spectacle plane using ETDRS letter charts. Trial lenses will be used to induce 1.0 D of astigmatism ATR, defined as -0.50/+1.00 D at approximately 90 degrees on the optical axis. VA will be measured in logMAR, with a lower logMAR value indicating better visual acuity. The change in VA before and after inducing astigmatism will be reported. One eye (first implanted eye) will be assessed. This is a co-primary endpoint.
Mean difference in monocular Distance Corrected Near Visual Acuity (DCNVA) (40 cm) before and after inducing 1.0 D astigmatism - ATR | Day 0, coinciding with IOL implantation at least 4 months prior to visit
  DCNVA will be assessed with distance correction in place (plus or minus power) at a distance of 40 cm from the spectacle plane using ETDRS letter charts. Trial lenses will be used to induce 1.0 D of astigmatism ATR, defined as -0.50/+1.00 D at approximately 90 degrees on the optical axis. VA will be measured in logMAR, with a lower logMAR value indicating better visual acuity. The change in VA before and after inducing astigmatism will be reported. One eye (first implanted eye) will be assessed. This is a co-primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Surgical CRD, Study Director — Alcon Research, LLC
Locations (3):
- United States (3):
  - Grosinger, Spigelman & Grey Eye Surgeons, P.C, Bloomfield Hills, Michigan
  - Key-Whitman Eye Center, Dallas, Texas
  - Berkeley Eye Center, Sugar Land, Texas